CLINICAL TRIAL: NCT04989985
Title: Perioperative SOX Plus Sintilimab Compared With Perioperative SOX in the Locally Advanced Esophagogastric Junction Adenocarcinoma: an Open-label, Phase 2 Randomised Controlled Trial
Brief Title: S-1 and Oxaliplatin (SOX) Plus Sintilimab in the Locally Advanced Esophagogastric Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Junsheng Peng, Chief, professor, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOLAR
Record Dates: First submitted 2021-06-16; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Locally Advanced Gastroesophageal Junction Adenocarcinoma; Chemotherapy Effect
Keywords: Locally Advanced Gastroesophageal Junction Adenocarcinoma; sinitilimab; SOX; peri-operative chemotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Comparator (Active Comparator): SOX: Oxaliplatin+S-1
  Oxaliplatin: 130mg/m2, iv drip for 2h, d1, q3w;
  S-1:40~60mg Bid, d1~14, q3w;
  Neoadjuvant chemotherapy for 2-4 cycles, adjuvant chemotherapy for 4-6 cycles.
  Interventions: Drug: Oxaliplatin+S-1
- Experimental (Experimental): Sinitlimab + SOX； SOX: Oxaliplatin+S-1
  Sinitlimab: 200mg, ivdrip, d1, q3w;
  Oxaliplatin: 130mg/m2, iv drip for 2h, d1, q3w;
  S-1:40~60mg Bid, d1~14, q3w;
  Neoadjuvant chemotherapy for 2-4 cycles, adjuvant chemotherapy for 4-6 cycles.
  Interventions: Drug: Sinitilimab+oxaliplatin+S-1

INTERVENTIONS:
Drug: Oxaliplatin+S-1 — Drug: Oxaliplatin Oxaliplatin: 130mg/m2，iv drip for 2h，d1, q3w
  Drug: S-1 S-1: 40~60mg Bid，d1~14, q3w
  Other Names: SOX
  Arms: Active Comparator
Drug: Sinitilimab+oxaliplatin+S-1 — Drug: Sintilimab Sintilimab, recombinant humanized anti-PD-1 monoclonal antibody for injection; 200mg ivdrip, d1, q3w.
  Other Name: PD-1 antibody
  Drug: Oxaliplatin Oxaliplatin: 130mg/m2，iv drip for 2h，d1, q3w
  Drug: S-1 S-1: 40~60mg Bid，d1~14, q3w
  Other Names: Sinitilimab+SOX
  Arms: Experimental

SUMMARY:
For locally advanced adenocarcinoma of esophagogastric junction(AEG) (cT3-4aN+M0), neoadjuvant chemotherapy was improved to downstage T and N stage, increase the resectability of tumor, and finally improve the long-term survival. Combination of perioperative PD-1 antibody and chemotherapy for locally advanced AEG could be a novel therapy to increase response rate and resectability and reduce recurrence rate. Sintilimab in this study is an anti-PD-1 monoclonal antibody for injection which has been approved for several malignant tumors. This study is a multi-center, open-label, randomized phase II clinical trial to evaluate tolerability, safety and efficacy of sintilimab in combination with perioperative chemotherapy in locally advanced AEG.

DETAILED DESCRIPTION:
Gastric cancer is one of the most common malignancies in China with incidence and mortality both ranking the 2nd among malignancies in China. Unfortunately, over 70% of gastric cancer patients in China were diagnosed in advanced stage, and more than 80% of adenocarcinoma of esophagogastric junction(AEG) were advanced stage. Locally advanced AEG (cT3-4aN+M0) could be cured by multi-disciplinary therapies including surgery, chemotherapy and radiotherapy. As proved, Neoadjuvant chemotherapy can downstage T and N stage, increase the resectability of tumor, and finally improve the long-term survival in AEG patients. However, the therapeutic effects remain unsatisfactory. PD-1 antibody has demonstrated its efficacy in metastatic AEG and has been proved to be effective in neoadjuvant setting in lung cancer and melanoma. Combination of perioperative PD-1 antibody and chemotherapy for locally advanced could be a novel therapy to increase response rate and resectability and reduce recurrence rate. Sinitilimab in this study is an anti-PD-1 monoclonal antibody for injection which has been approved for lymphoma. This study is a multi-center, open-label, randomized phase II clinical trial to evaluate tolerability, safety and efficacy of sinitilimab in combination with perioperative chemotherapy（SOX: oxaliplatin plus S-1） in locally advanced AEG.

ELIGIBILITY:
Inclusion Criteria:

1. Written (signed) informed consent;
2. Histologically CT/MRI confirmed cT3-4aN+M0 Esophagogastric Junction Adenocarcinoma;
3. Consent to send tumor tissue from biopsy or resection for PD-L1, EBV, MSI detection;
4. Female or male, 18-75 years;
5. ECOG 0-1, no surgery contraindications;
6. Physical condition and adequate organ function to ensure the success of abdominal and/or thoracic surgery;
7. Expected survival ≥ 6 months;
8. Adequate hematological, liver, renal and coagulation function; 1) Platelet (PLT) count ≥100,000 /mm3; 2) White Blood cell（WBC）count ≥4,000 /mm3 and ≤15,000 /mm3 ；Neutrophil count (ANC) ≥1,500 /mm3; 3) Hemoglobin (Hb) level ≥9.0 g/dl; 4) International normalized ratio (INR) ≤1.5; 5) Prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤1.5×ULN; 6) Glycosylated hemoglobin (HbA1c) <7.5%; 7) Total bilirubin (TBIL) level ≤1.5×ULN; 8) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) level ≤2.5×ULN (≤5×ULN in case of liver metastasis); 9) Alkaline phosphatase level ≤2.5×ULN (≤5×ULN in case of liver metastasis); 10) Serum creatinine (Cr) level ≤1.5×ULN and creatinine clearance ≥60 ml/min;
9. Patients with Good compliance, who can cooperate with the laboratory, auxiliary examinations and corresponding specimen collection of this program set;
10. Females of child bearing age must have a negative pregnancy test, and have to take contraception measures and avoid breast feeding during the study and for 6 months after the last dose; male subjects must agree to taken contraception measures during the study and for 6 months after the last dose.

Exclusion Criteria:

1. Suffer from other active malignant tumors within 5 years or at the same time. Cured localized tumors, such as skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, prostate carcinoma in situ, cervical carcinoma in situ, breast carcinoma in situ, etc. can be included in the group.
2. Patients who are planning to undergo or have previously received organ or bone marrow transplantation.
3. Myocardial infarction or poorly controlled arrhythmia (including QTc interval ≥ 450 ms for males and ≥ 470 ms for females) occurred within 6 months before the first medication (QTc interval is calculated by Fridericia's formula).
4. There is NYHA standard grade III to IV cardiac insufficiency or color Doppler ultrasound examination: LVEF (left ventricular ejection fraction) <50%.
5. Human immunodeficiency virus (HIV) infection.
6. Suffer from active tuberculosis.
7. Past and present patients who have interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severely impaired lung function, etc., which may interfere with the detection and management of suspected drug-related lung toxicity.
8. There is a known active or suspicious autoimmune disease. Except those who were in a stable state of the disease at the time of enrollment (no need for systemic immunosuppressive therapy).
9. Received treatment with live vaccine within 28 days before the first administration; except for the treatment of seasonal influenza with inactivated viral vaccine.
10. Patients who need to receive systemic corticosteroids (> 10 mg/day curative dose of prednisone) or other immunosuppressive drugs within 14 days before the first medication or during the study period. However, the following conditions are allowed to enter the group: in the absence of active autoimmune diseases, patients are allowed to use topical or inhaled steroids, or adrenal hormone replacement therapy with a dose of ≤ 10 mg/day prednisone.
11. Any active infection that requires systemic anti-infective treatment occurs within 14 days before the first administration of the drug; except for receiving preventive antibiotic treatment (such as prevention of urinary tract infection or chronic obstructive pulmonary disease).
12. Have received other antibody/drug treatments for immune checkpoints in the past, such as PD-1, PD-L1, CTLA4 and other treatments.
13. Are receiving other clinical research treatments, or the planned start of this research treatment is less than 14 days from the end of the previous clinical research treatment.
14. Known to have a history of severe allergies to any monoclonal antibodies or study drug excipients.
15. Known history of psychotropic drug abuse or drug use; patients who have stopped drinking can be included in the group.
16. There are patients who may increase the risk of participating in research and research medication, or other severe, acute and chronic diseases, who are not suitable for participating in clinical research based on the judgment of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
pCR | From the initiation date of first cycle (each cycle is 21 days) to the date of operation, an average of 12 weeks.
  pathological complete response rate

SECONDARY OUTCOMES:
TRG0/1 | From the initiation date of first cycle (each cycle is 21 days) to the date of operation, an average of 12 weeks.
  Pathological tumor regression grade 0/1
R0 resection rate | rom the initiation date of first cycle (each cycle is 21 days) to the date of operation, an average of 12 weeks.
  Rate of microscopically margin-negative resection
DFS | From the initiation date of first cycle (each cycle is 21 days) to the date of first documented symptoms of cancer, assessed up to 3 years
  the length of time after primary treatment for a cancer ends that the patient survives without any signs or symptoms of that cancer.
RFS | From the initiation date of first cycle (each cycle is 21 days) to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  The Kaplan-Meier survival from the initiation date of first cycle until the date of first documented recurrence
OS | From the initiation date of first cycle (each cycle is 21 days) to the date of death from any cause, whichever came first, assessed up to 5 years
  The Kaplan-Meier survival from the initiation date of first cycle until death from any cause or the last follow-up date.

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Sheng Peng, Dr, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The sixth affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China